CLINICAL TRIAL: NCT02749825
Title: A Multicenter, Randomized Clinical Investigation of Trelstar Versus Continued Therapy in Patients Receiving Lupron or Zoladex for Advanced Prostate Cancer
Brief Title: Comparison of Trelstar Versus Lupron or Zoladex in Advanced Prostate Cancer
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Withdrawal of funding support
Sponsor: Pharmatech (Industry)
Collaborators: Manyak, Michael, M.D. (Individual); Watson Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUI-02809
Record Dates: First submitted 2012-05-08; First posted 2016-04-25 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2012-05

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Trelstar
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Triptorelin Pamoate; Leuprolide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Trelstar (Experimental): Per prescribing information
  Interventions: Drug: Trelstar
- Lupron (Active Comparator): Per prescribing information
  Interventions: Drug: Lupron
- Zoladex (Active Comparator): Per prescribing information
  Interventions: Drug: Zoladex

INTERVENTIONS:
Drug: Trelstar — As labeled
  Other Names: Triptorelin pamoate
  Arms: Trelstar
Drug: Lupron — As labeled
  Other Names: luprolide acetate for depot suspension
  Arms: Lupron
Drug: Zoladex — As labeled
  Other Names: goserelin acetate
  Arms: Zoladex

SUMMARY:
This research study looks at Testosterone levels in patients receiving Trelstar versus those receiving Lupron or Zoladex. These drugs have been approved for treatment of Prostate Cancer by the FDA.

DETAILED DESCRIPTION:
Patients who are currently receiving Lupron or Zoladex will be consented and then randomized to receive either continued treatment with the drug they have been on, or will be randomized to Trelstar for a period of 3 months. At the end of that period, testosterone and prostate serum antigen (PSA) levels will be drawn and compared to their previous levels to determine if Trelstar is as effective as the previous treatment.

ELIGIBILITY:
Inclusion Criteria:

* Advanced Prostate Cancer
* Currently taking Lupron or Zoladex
* Stable PSA
* Baseline testosterone below castration level
* Life expectancy > 6 months
* Eastern Cooperative Oncology Group performance status of 0-2
* Signed, approved informed consent.

Exclusion Criteria:

* Known hypersensitivity to any leuteinizing hormone releasing hormone (LHRH) agonist
* Ongoing therapy with hyperprolactinemic agents
* Antiandrogen therapy within 28 days prior to study start
* Prior Orchiectomy, hypophysectomy or adrenalectomy
* Chemotherapy, radiotherapy, or prostatectomy within 28 days prior to study start
* Use of any investigational agent 3 months prior to enrollment
* Use of systemic corticosteroids within 28 days or during study
* Other malignancies within 2 yrs prior to study start, except curatively treated skin cancers
* Severe kidney or liver failure, based on adequate lab values
* Other medical conditions which would be likely to interfere with compliance or completion of study requirements

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2002-09; Primary Completion 2006-05 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
Maintenance of serum testosterone at or below castration level (50ng/dL) | 12 weeks
  Primary efficacy

SECONDARY OUTCOMES:
Serum testosterone level at end of study | Week 12
  Secondary efficacy
Change in serum testosterone from baseline to end of study | Baseline and week 12
  Secondary efficacy
Incidence and severity of adverse events | 12 weeks
  Treatment tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Michael Michael Manyak, MD, Principal Investigator — Georege Washington University
Locations (11):
- United States (11):
  - Arizona Urologic Specialists, Tucson, Arizona
  - Heritage Physician Group - Urology Department, Hot Springs, Arkansas
  - California Oncology of the Central Valley, Fresno, California
  - San Bernardino Urological Associates Medical Group, San Bernardino, California
  - UroSearch, Ocala, Florida
  - Scott A Slavis, MD, PC, Las Vegas, Nevada
  - Shaukat M Qureshi, MD, Pennsville, New Jersey
  - Brooklyn Heights Urology Associates, Brooklyn, New York
  - Jazrawi-Atallah, P.C., Brooklyn, New York
  - Albemarle Urology Clinic, PA, Albemarle, North Carolina
  - Raj P. Chopra MD, PC, Bloomsburg, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Pharmatech - The Research Link website — http://www.pharmatech.com